CLINICAL TRIAL: NCT05866432
Title: Phase II Study of Datopotamab-Deruxtecan (Dato-DXd; DS-1026a) in Triple-negative Breast Cancer Patients With Newly Diagnosed or Progressing Brain Metastases
Brief Title: Phase II Study of Dato-DXd in Triple-negative Breast Cancer Patients With Newly Diagnosed or Progressing Brain Metastases
Acronym: TUXEDO-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Rupert Bartsch, Assoc.-Prof. PD Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUXEDO-2
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Datopotamab-deruxtecan (Experimental): Datopotamab-deruxtecan (DS-1062a) 6.0 mg/kg body weight i.v. on day 1 once every three weeks
  Interventions: Drug: Datopotamab deruxtecan

INTERVENTIONS:
Drug: Datopotamab deruxtecan — Will be given until PD or withdraw
  Other Names: S-1062a

SUMMARY:
Datopotamab-deruxtecan in triple-negative breast cancer patients with newly diagnosed or progressing brain metastases.

DETAILED DESCRIPTION:
Datopotamab-deruxtecan will be administered at a dose of 6.0 mg/kg body weight i.v. on day

1 once every three weeks in triple-negative breast cancer patients with newly diagnosed or progressing brain metastases. Response rate by RANO-BM criteria is definied as primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer
* Triple-negative disease as defined by immunohistochemistry (IHC) and/or c-erb-B2 gene amplification status. For the definition of hormone-receptor negative disease, a cut-off of <10% tumour cells with positive staining of oestrogen- and progresteron-receptors is required
* Newly diagnosed untreated brain metastases or brain metastases progressing after prior local therapy
* Measurable disease (RANO-BM criteria)
* No indication for immediate local treatment
* Accompanying type II leptomeningeal disease allowed (suspected LMD by clinical findings and neuroimaging)
* KPS ≥70%, ECOG ≤2 Indication for systemic anti-cancer treatment
* Prior exposure to PD-1, PD-L1 inhibitors and TROP-2 targeted agents allowed
* Life expectancy of at least 3 months
* Age ≥18 years
* Patient must be able to tolerate therapy
* Adequate bone-marrow, liver and kidney function
* Adequate treatment washout period before enrolment, defined as:
* Major Surgery: ≥3 weeks
* Radiation therapy to the chest: ≥4 weeks
* Palliative radiation therapy to other areas: ≥2 weeks
* Chemotherapy, small-molecule targeted agents: ≥3 weeks
* Antibody-based treatment: ≥4 weeks (concurrent therapy with denosumab allowed)
* Patient must be capable of understanding the purpose of the study and have given written informed consent

Exclusion Criteria:

* Known hypersensitivity to Dato-DXd or any of the drug components
* Use of any investigational agent within 28 days prior to initiation of treatment
* History of malignancies other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 3 years including contralateral breast cancer
* Other anticancer therapy, including cytotoxic, targeted agents, immunotherapy, antibody, retinoid, or anti-cancer hormonal treatment with the exception of osteoprotective therapies such as denosumab or bisphosphonates
* Concomitant radiotherapy
* A history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), left ventricular ejection fraction <50%, arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities, and long QT syndrome (QTc interval >470 ms)
* Inadequate bone marrow function at baseline prior to study entry
* Inadequate kidney function
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease including active or uncontrolled infections with hepatitis B and C
* Participants with known hepatitis B and C are eligible if they:

  1. Have been curatively treated for HCV infection as demonstrated clinically and by viral serologies
  2. Have received HBV vaccination with only anti-HBs positivity and no clinical signs of hepatitis
  3. Are HBsAg- and anti-HBc+ (i.e., those who have cleared HBV after infection) and meet conditions i-iii below:
  4. Are HBsAg+ with chronic HBV infection (lasting 6 months or longer) and meet conditions 1-3 below:
  5. HBV DNA viral load <2000 IU/mL
  6. Have normal transaminase values, or, if liver metastases are present, abnormal transaminases, with a result of AST/ALT <3 × ULN, which are not attributable to HBV infection
  7. Start or maintain antiviral treatment
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Has a history of non-infectious ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
* Subjects with bronchopulmonary disorders who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study
* Patients with active opportunistic infections
* Known human immunodeficiency virus (HIV) infection that is not well controlled
* Pregnant or lactating women
* Women with childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy.
* Male subjects unable or unwilling to use adequate contraception methods
* Patients with known substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results
* Patients requiring concomitant use of chronic systemic (IV or oral) corticosteroids at doses higher than 8 mg dexamethasone per day or other immunosuppressive medications except for managing adverse events; (inhaled steroids or intra articular steroid injections are permitted in this study)
* Patients with significant corneal disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Intracranial response rate to datopotamab-deruxtecan | From date of inclusion until the date of firstdocumented progression or date of death from any cause or treatmentdiscontinuation from any other reason, whichever came first, assessedup to 36 months]
  Measured according to RANO-BM criteria

SECONDARY OUTCOMES:
Entracranial response rate to datopotamab-deruxtecan | From date of inclusion until the date of firstdocumented progression or date of death from any cause or treatmentdiscontinuation from any other reason, whichever came first, assessedup to 36 months]
  Measured according to RECIST 14.1 criteria
Progression-free survival | From date of inclusion until the date of firstdocumented progression or date of death from any cause or treatmentdiscontinuation from any other reason, whichever came first, assessedup to 36 months]
  Time from inclusion until progression
Overall Survival | From date of inclusion until the date of firstdocumented progression or date of death from any cause or treatmentdiscontinuation from any other reason, whichever came first, assessedup to 36 months]
  Time from inclusion until progression
Safety & tolerability of datopotamab-deruxtecan in terms of haematologic and non-haematologic side effect | From date of inclusion until the date of firstdocumented progression or date of death from any cause or treatmentdiscontinuation from any other reason, whichever came first, assessedup to 36 months]
  Assessment of clinical adverse events & laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Rupert, MD, Principal Investigator — Medical University Vienna
Locations (1):
- AKH Universitaetsklinikum Vienna, Department f. Internal medicine I, oncology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No